CLINICAL TRIAL: NCT02383056
Title: Doubleblinded, Randomized, Controlled Trial to Study the Effect of Omnilux Light Emitting Diode on Wound Healing Following Lower Extremity Surgical Wounds Left to Heal by Second Intention
Brief Title: Doubleblinded RCT of the Omnilux on Lower Extremity Surgical Wounds Left to Heal by Second Intention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sufficient enrollment achieved for outcome measures
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Keyvan Nouri, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20120475
Record Dates: First submitted 2015-02-27; First posted 2015-03-09 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Wound
Keywords: wound; secondary intention healing; lower extremity
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Group (Group 1) (Sham Comparator): This group will receive 4 sessions of Omnilux sham light, starting 1 week after the surgery. Frequency: 1 session every week (+/- 3 days), for 4 weeks. Session duration: 20 minutes
  Interventions: Device: Omnilux Sham
- Treatment group (Group 2) (Experimental): This group will receive 4 treatment sessions with Omnilux 633nm LED, starting 1 week after the surgery. Frequency: 1 session every week (+/- 3 days), for 4 weeks. Session duration: 20 minutes
  Interventions: Device: Omnilux

INTERVENTIONS:
Device: Omnilux — Photomodulation irradiated with a 633 +/- 3 mm light source for 20 minutes (105 mW/cm, 126 J/cm)
  Arms: Treatment group (Group 2)
Device: Omnilux Sham — Sham light instead of phototherapy from the same light device
  Arms: Sham Group (Group 1)

SUMMARY:
The goal of the study is to evaluate the effectiveness of the light-emitting diode (LED) in promoting healing of the wound on lower leg as a result of surgery. Wounds on the lower leg heal more slowly than wounds on the head and neck; they can also remain deep red for six months to one year. Doctors usually allow a lower leg surgical wound to heal by itself, without stitches or other additional treatment. This is because leg wounds do not hold stitches well and stitches could cause other problems. A major drawback of allowing a surgical wound on the lower leg to heal by itself is the long healing time that can often take months. The investigators wish to evaluate if the LED light treatment of the surgical wound will improve the healing of your wound.

In order to test if leg wounds heal faster after treatment with LED, half of the patients in the study will receive the LED (Group 2) and half will not receive treatment with LED but will receive a "sham light" treatment (Group 1). Essentially, a sham light treatment refers to regular light (not LED) exposure for 20 minutes. The sham light comes from the same device as the treatment light (Omnilux machine) however, this light has no anticipated effects on wound healing and is used simply to reduce the amount of bias that sometimes complicates the results of these studies. There is no added risk or benefit for the patients in the control group exposed to the sham light. Both groups will receive the standard care of wounds on the lower extremity.

DETAILED DESCRIPTION:
Group 2 of this study will receive the LED and half will not receive treatment with LED but will receive a "sham light" treatment (Group 1). Essentially, a sham light treatment refers to regular light (not LED) exposure for 20 minutes. The sham light comes from the same device as the treatment light (Omnilux machine) however, this light has no anticipated effects on wound healing and is used simply to reduce the amount of bias that sometimes complicates the results of these studies. There is no added risk or benefit for the patients in the control group exposed to the sham light. Both groups will receive the standard care of wounds on the lower extremity.

Groups 1 and 2 will receive 4 sham light or treatment sessions, respectively (one session every week for 4 weeks). After these sessions are done, all subjects will continue weekly follow up visits until the wound is closed, or 3 months after the surgery have passed; which ever happens first.

One final follow up visit will occur 1 week after the wound closed.

ELIGIBILITY:
Inclusion Criteria:

* Surgical defect on the lower extremity left to heal by secondary intention.
* If women of child bearing potential, contraceptive measures should be used
* Maximum size of wound is 5cm x5cm; there is no minimum size for the wound.

Exclusion Criteria:

* History of porphyria photosensitive eruptions, diabetes mellitus, history of venous insufficiency, known history of peripheral arterial disease (ABI <0.8)
* Use of any ointments or creams containing photosensitizers (coumarins or porphyrins) should be discontinued for 2 weeks prior
* Use of systemic or local retinoids for the past 6 months.
* Current pregnancy or breastfeeding
* History of metastatic cancer.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Nouri, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospital and Clinics/Sylvester Comprehensive Cancer Center, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Group (Group 1): This group will receive 4 sessions of Omnilux sham light, starting 1 week after the surgery. Frequency: 1 session every week (+/- 3 days), for 4 weeks. Session duration: 20 minutes
  Omnilux sham light
- Treatment Group (Group 2): This group will receive 4 treatment sessions with Omnilux 633nm LED, starting 1 week after the surgery. Frequency: 1 session every week (+/- 3 days), for 4 weeks. Session duration: 20 minutes
  Omnilux: 633nm
Period: Overall Study
Arm/Group | Sham Group (Group 1) | Treatment Group (Group 2)
Started | 7 | 7
Completed | 6 | 5
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Group (Group 1) | Treatment Group (Group 2) | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (7.39) | 72.6 (5.41) | 71.0 (6.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Required for the Wound to Heal Completely
Description: Assessment by the physician indicating wound closure
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sham Group (Group 1) | Treatment Group (Group 2)
Number analyzed (Participants) | 6 | 5
days | 48.67 (11.10) | 63.20 (12.20)

2. Secondary Outcome: Change in Relative Area of the Surgical Wound Remaining
Description: Initial area * ((total area in the evaluated week/total area in the first week) * 100) and reported as a percentage (%)
Time Frame: Week 1 to Week 2, Week 2 to Week 3, Week 3 to Week 4
Measure: Mean (Standard Deviation); unit: Percentage of Wound Remaining
Arm/Group | Sham Group (Group 1) | Treatment Group (Group 2)
Number analyzed (Participants) | 6 | 5
Percentage of Wound Remaining
  Week 1 to Week 2 | 90.80 (19.40) | 96.0 (23.70)
  Week 2 to Week 3 | 60.70 (8.71) | 77.40 (5.76)
  Week 3 to Week 4 | 53.10 (17.0) | 45.98 (20.5)

3. Secondary Outcome: Change in Total Surface Area of the Surgical Wound
Description: A blinded investigator manually outlines the wound using a digital planimetry device to measure the surface area in square centimeters.
Time Frame: Week 1 to Week 2, Week 2 to Week 3, Week 3 to Week 4, Week 1 to Week 4
Measure: Mean (Standard Deviation); unit: Cm^2
Arm/Group | Sham Group (Group 1) | Treatment Group (Group 2)
Number analyzed (Participants) | 6 | 5
Cm^2
  Week 1 to Week 2 | -0.18 (0.57) | -0.25 (0.62)
  Week 2 to Week 3 | -0.93 (0.82) | -0.48 (0.44)
  Week 3 to Week 4 | -0.27 (0.60) | -0.80 (0.34)
  Week 1 to Week 4 | -1.38 (1.03) | -1.53 (0.12)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Sham Group (Group 1) | Treatment Group (Group 2)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 3/7 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Group (Group 1) (N=7) | Treatment Group (Group 2) (N=7)
Erythema (Skin and subcutaneous tissue disorders) | 3 | 5
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Tenderness (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT02383056/Prot_SAP_000.pdf